CLINICAL TRIAL: NCT00277849
Title: Collection of Blood From Persons With Hemoglobin and Erythrocyte Polymorphisms for Laboratory Malaria Research
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060074; 06-I-0074
Record Dates: First submitted 2006-01-14; First posted 2006-01-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-07-20

CONDITIONS: Hemoglobin Mutations; Erythrocyte Variants
Keywords: Sickle; Hemoglobinopathy; Thalassemia; G6PD; Plasmodium; Erythrocyte Variant; Hemoglobin Variant; Healthy Volunteer; HV
MeSH Terms: conditions — Hemoglobinopathies; Thalassemia; Malaria

SUMMARY:
This study will collect blood samples for use in laboratory studies of malaria. The World Health Organization reports that 40 percent of the world's population is at risk for malaria, mostly in the poorest countries. It is a serious disease caused by parasites. Each year, 300-500 million infections lead to more than a million deaths. However, there are traits in red blood cells (erythrocyte) that protect people against malaria. In this study, polymorphism refers to the various kinds of red blood cell traits.

The sickle cell trait is an example of one that seems to offer a natural survival advantage in children where malaria is common. Researchers at the Laboratory of Malaria and Vector Research are investigating ways in which the blood cell traits can offer such protection, and new knowledge gained can bring about medical advances. Of particular importance is studying how the malaria organism, Plasmodium, survives inside different red blood cells. A steady, consistent, and reliable supply of fresh whole blood is necessary for testing.

Patients 18 to 65, weighing more than 110 lbs. and who do not have anemia or known HIV, Hepatitis C, or Hepatitis B may be eligible for this study.

Patients will undergo a medical history and general assessment including vital signs of temperature, heart rate, and blood pressure. Blood will be collected from a vein in the arm, or rarely a vein in the hand. A complete blood count, or CBC, will be done to ensure that blood levels are sufficient and that blood donation is safe for a patient to do. Patients need to have enough hemoglobin, the part of red blood cells that transports oxygen throughout the body. The blood will also be tested to confirm the type of red blood cell traits of patients. About 1 to 8 tablespoons may be collected, but most blood samples will be small, that is, 1 to 4 teaspoons. After the patients' first visit, sessions will take 5-20 minutes. Blood collection will total no more than 2 cups from a donor during any 6-week period. Although the frequency of blood donations is not known at this time, it is unlikely that a patient will be asked to donate blood more than four times a year. It may be important for patients to undergo a repeat CBC or tests for blood chemistry if results are needed for research. Risks associated with blood collection are considered minimal. They include discomfort, occasional bruising or bleeding at the puncture site, and faintness.

In this study, it is possible that a small amount of blood may be stored for future research, to help the researchers to learn more about malaria. There are no plans for the results from the various research laboratory tests to be made available to patients or to their private doctors. However, patients in this study may discuss the results of routine medical tests with the study investigators. Some of the blood collected will be tested for genetic conditions. Through genetic testing, researchers can learn more about how health or illness may be passed on to people by their parents, or from people to their children. All results of tests will remain confidential. Blood samples will be labeled by code, and reference to patients' identities will be protected.

Participants will receive $50 for each blood donation. This study will not have a direct benefit for participants. Future research that uses their blood samples will help researchers to learn about malaria as well as how to prevent or treat the disease.

DETAILED DESCRIPTION:
This protocol is designed to provide a mechanism for investigators in the Laboratory of Malaria and Vector Research (LMVR) to collect and process peripheral blood samples from volunteer donors. Donors who meet standard eligibility criteria will be recruited to donate blood via standard phlebotomy techniques at the NIH Clinical Center.

The LMVR has ongoing in vitro studies to characterize the effects of hemoglobin mutations and erythrocyte polymorphisms on the pathogenesis of Plasmodium falciparum, the agent of the most deadly malaria in humans. G6PD deficiency, hemoglobinopathies such as HbS, HbC, and HbE, and the thalassemias are thought to have evolved as protective traits against malaria in endemic areas of the world. However, the mechanisms by which these mutations exert their protective influence are largely unknown. Culturing P. falciparum in erythrocytes carrying protective traits will allow researchers in LMVR to characterize the cellular and molecular bases of protection using in vitro methods such as growth analyses and electron microscopy. To this effect, patients with known or suspected erythrocyte variants will be recruited in addition to normal controls.

Signed informed consent will be obtained by an authorized investigator. The nature of the study as well as the risks and benefits of the donation process will be explained to each participant. Donors will be compensated for each blood donation or for unsuccessful attempts at venipuncture. Samples will be used solely for in vitro research. To ensure confidentiality, blood will be assigned a unique code; investigators listed on this protocol will serve as the custodians of the codes that link the samples to the donors' identities.

ELIGIBILITY:
* INCLUSION CRITERIA:

Normal volunteer or volunteer with a known or suspected erythrocyte mutation.

Age greater than or equal to 18 and less than or equal to 65 years old.

Weight greater than 110 pounds.

Ability to sign the consent form.

Willingness to comply with study procedures.

EXCLUSION CRITERIA:

Transfusion of any blood products within the past 90 days.

Active bleeding.

Clinically apparent and/or symptomatic anemia (pallor, orthostasis, etc).

Self-reported history of HIV, Hepatitis B virus, or Hepatitis C virus infection.

Severe chronic disease (e.g. end-stage renal failure, malignancy, etc).

Significant medical history, physical examination, or laboratory test results indicating that the subject should not participate in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2006-01-11; Study Completion 2010-07-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States